CLINICAL TRIAL: NCT03529994
Title: Work of Breathing and Oxygen Saturation Stability in Infants With Respiratory Insufficiency While Receiving Various Flow Rates of High Flow Nasal Cannula
Brief Title: Work of Breathing and Oxygen Saturation in Infants Receiving High Flow Nasal Cannula (HFNC)
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other)
Responsible Party: Sponsor
Other Study IDs: DDD603875
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-05

CONDITIONS: High Flow Nasal Cannula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrollment
  Interventions: Other: Enrollment

INTERVENTIONS:
Other: Enrollment — All infants enrolled will have work of breathing assessed.

SUMMARY:
The purpose of this study is to compare work of breathing on different levels of high flow respiratory support on infants born between 27 and 37 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 27 and 37 weeks corrected gestational age
* >4 days PNA
* Stable (i.e. not meeting exclusion criteria) and receiving non-invasive respiratory support (HFNC) for ≥ 12 hours
* Requiring ≤ 40% supplemental FiO2 as determined by the clinical care team for clinical care purposes independent of this study

Exclusion Criteria:

* Infants with skeletal, neuromuscular, or abdominal surgical disorders that affect the accuracy of WOB measurements

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Convenience sample of infants on HFNC admitted to our NICU who meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Work of breathing indices | 2 hours
  Altering HFNC flow rates and its effect on work of breathing indices in preterm infants with respiratory insufficiency.

SECONDARY OUTCOMES:
Intermittent hypoxia | 2 hours
  Altering HFNC flow rates and its effect on intermittent hypoxia in preterm infants with respiratory insufficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Kovatis, MD, Principal Investigator — Christiana Care Health Services, Inc.
Locations (1):
- Christiana Care Health Services, Inc., Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No